CLINICAL TRIAL: NCT00203567
Title: Carbamazepine Extended-Release for the Treatment of Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: Shire (Industry)
Responsible Party: Lori L. Davis, M.D.; Chief, Research Service, Tuscaloosa Research Education & Advancement Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREAC Equetro in Bipolar; TREAC Equetro in Bipolar
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Bipolar Depression
Keywords: bipolar depression; carbamazepine ER; Equetro
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Equetro (Active Comparator): Equetro
  Interventions: Drug: carbamazepine ER

INTERVENTIONS:
Drug: carbamazepine ER — Active study drug, no comparator

SUMMARY:
To study the efficacy and safety of beaded extended-release Carbamazepine (Equetro) in the treatment of patients with Bipolar Disorder with a Major Depressive Episode.

DETAILED DESCRIPTION:
Patients with Bipolar I or II Disorder with a Major Depressive Episode who sign informed consent and meet eligibility criteria will begin treatment with extended release carbamazepine (ERC-CBZ ). The dose of ERC-CBZ will be initiated at 200mg twice daily and increased as tolerated by 200mg/day every 3 days up to 1200mg/day by week 2 (target dose). Then the dose may be increased at the investigator's discretion, up to1600mg/day as tolerated by week 8, if needed for a greater therapeutic response. Efficacy will be assessed biweekly with the Montgomery-Asberg Depression Rating Scale (MADRS) and Clinical Global Impression-Bipolar (CGI-BP). Safety is assessed biweekly with adverse events self-reports and laboratory evaluations. ).

ELIGIBILITY:
Inclusion Criteria:

* Age 19 -65.
* Diagnosis of Bipolar I or II Disorder, currently experiencing a major depressive episode without psychotic features, as confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I.).
* Must have experienced at least two previous mood episodes during the past 10 years, at least one of which was a hypomanic, full manic or mixed episode. The current depressive episode must be ≥ 2 weeks, but ≤ 2 years in duration.
* Must currently have clinically significant depressive symptoms as defined by a CGI-S total score of ≥ 4.
* Must have been washed out of all psychotropic medications (except for the allowed concomitant sedatives for insomnia) for their bipolar illness for at least 3 days for mood stabilizers and 1 week for antidepressants prior to study drug initiation (medications should be tapered at the investigator's discretion prior to washout), while continuing to meet entry criteria for depressive symptoms. Must be willing to discontinue all psychotropic medication (except for the allowed concomitant sedative for insomnia) during the study period.
* No substance abuse/dependence for the previous 4 weeks (except for nicotine/caffeine)
* Must give informed consent, and/or consent must be obtained from a legally acceptable representative (as required by IRB) prior to the initiation of any protocol required procedures.
* Must be able to understand the nature of the study, agree to comply with the prescribed dosage regiments, report for regularly scheduled office visits and communicate to study personnel about adverse events and concomitant medication.
* Women of childbearing potential (WOCBP) must use medically approved methods of birth control to avoid pregnancy throughout the study and for up to four weeks after completion of the study in such a manner that the risk of pregnancy is minimized. WOCBP must have a negative serum or urine pregnancy test within 72 hours prior to the start of the study.
* Male or female, any race or ethic origin

Exclusion Criteria:

* Patients with current diagnosis of delirium, dementia, amnestic or other cognitive disorder; schizophrenia; borderline or antisocial personality disorder; or any other mental disorder that would interfere with efficacy or safety evaluations or compliance.
* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to four weeks after completion of the study. Acceptable methods include oral, injectable or implanted contraceptives, intrauterine devices or barrier methods such as condoms, diaphragm, and spermicides. Women who are pregnant or breast-feeding, or who plan to become pregnant during the study.
* Patients at significant risk of committing suicide or homicide based on history, mental status exam, or investigator's judgment.
* Patients receiving psychotherapy (individual, group, marriage, or family therapy) unless participation has been regular for at least 3 months prior to randomization.
* Patients with clinically significant thyroid pathology that would interfere with efficacy or safety evaluations and patients with a thyroid stimulating hormone (TSH) level > 60% above the upper limit of normal. Patients who are undergoing treatment for their thyroid pathology (e.g. thyroid supplementation) should be stable for at least two months prior to randomization.
* Patients who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial, including but not limited to hepatic, renal respiratory, cardiovascular, endocrine, neurologic, or hematologic disease as determined by the clinical judgment of the investigator.
* Patients with a history of seizures (except for a single childhood febrile seizure, posttraumatic, alcohol withdrawal) or a history of severe head trauma, or stroke.
* Patients on medications that may have serious drug-drug interactions with ERC-CBZ
* Clinically significant abnormal laboratory tests results:

  * Platelets < 75,000/mm³
  * Hemoglobin < 9g/dL
  * Neutrophils, Absolute < 1000/mm³
  * SGOT (AST) >3x Upper limit of Normal
  * SGPT (ALT) > 3x Upper Limit of Normal
  * Creatinine >2mg/dL
  * Diastolic blood pressure >105 mmHg
  * TSH > 60% above Upper Limit of Normal
  * Detectable levels of cocaine and amphetamines in the urine drug screen.
  * Other abnormal laboratory test or vital sign result that in the investigator's judgment, is medically significant, in that it would impact the safety of the patient or the interpretation of the results.
* Patients who are known to be allergic or hypersensitivity to carbamazepine (or alternative formulations).
* Patients who have failed an adequate trial of carbamazepine (or alternative formulations) for bipolar depression.
* Patients who have had recent treatment with a long-acting antipsychotic in which the last dose was less than one full cycle plus one week
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g. infectious disease) illness during the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-08; Primary Completion 2007-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To study the efficacy and safety of beaded extended-release Carbamazepine (Equetro) in the treatment of patients with Bipolar Disorder with a Major Depressive Episode. | 8 weeks

SECONDARY OUTCOMES:
The treatment phase will include Mean Change from Baseline to Endpoint (Week 8 LOCF) on the CGI-BP, Q-LES-Q, and Ham-A. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (1):
- Tuscaloosa Research and Education Advancement Corporation, Tuscaloosa, Alabama, United States

REFERENCES:
- [Background] Swainston Harrison T, Keating GM. Extended-release carbamazepine capsules : in bipolar I disorder. CNS Drugs. 2005;19(8):709-16. doi: 10.2165/00023210-200519080-00006. PMID 16097852